CLINICAL TRIAL: NCT03339739
Title: Effects of Mandibular Exercises Effect in Pain Perception and Sensitivity in Women With Myofascial Pain, a Double Blind Randomized Clinical Trial.
Brief Title: Effects of Mandibular Exercises Effect on Pain Perception and Sensitivity in Mandibular Myofascial Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional Andres Bello (Other)
Responsible Party: Principal Investigator, Juan Fernando Oyarzo, Orofacial Pain & TMD Professor, Universidad Nacional Andres Bello
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PROPRGFO_2013/004
Record Dates: First submitted 2017-10-31; First posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Temporomandibular Disorders
Keywords: Musculoskeletal Pain; Orofacial Pain; Physical Therapy Modalities; Oral Contraceptives; Mandibular Diseases; Muscular Diseases; Risk factors; Contraceptive Usage; Pain, Chronic; Craniomandibular Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders; Musculoskeletal Pain; Facial Pain; Mandibular Diseases; Muscular Diseases; Contraception Behavior; Chronic Pain; Craniomandibular Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Isometric exercise Group (Experimental): Group of participants which perform Isometric mandibular exercises, once a day, for 21 days
  Interventions: Other: Isometric mandibular exercises
- Isotonic exercise Group (Active Comparator): Group of participants which perform Isotonic mandibular exercises, once a day, for 21 days
  Interventions: Other: Isotonic mandibular exercises
- Counseling Group (Placebo Comparator): Group of participants which receive education brochure and no further interventions.
  Interventions: Behavioral: Counseling group

INTERVENTIONS:
Other: Isometric mandibular exercises — daily video guided three-minutes routine in 21 days (days of OC consumption) of soft clenching over three millimeters silicone bars bilaterally on molars
  Arms: Isometric exercise Group
Other: Isotonic mandibular exercises — daily video guided three-minutes routine in 21 days (days of OC consumption) of isotonic dynamic contraction over calibrated cloth pegs on central incisors
  Arms: Isotonic exercise Group
Behavioral: Counseling group — subjects included in this group get an education brochure about the disorder and receive no further interventions
  Arms: Counseling Group

SUMMARY:
The effectiveness of mandibular exercises as a treatment of muscular Orofacial Pain is yet unknown. This study hypothesized that training exercises can be an effective therapy improving pain perception.

DETAILED DESCRIPTION:
Temporomandibular disorders (TMDs) represent heterogeneous musculoskeletal disorders, where most common presentation is mandibular muscle pain, which is also more common among female than men. Many interventions have been proposed for this pain control, regarding drugs, oral splints, relaxing exercises and self awareness but little is known about mandibular active contraction exercises. The aim of this study is to evaluate the effects of mandibular exercises in pain perception and sensitivity in women. A double blind randomized clinical trial will be conducted among fertile university student women with Oral Contraceptives (OC) use -to control hormonal influences-, with report of facial pain and myofascial pain diagnosis (RDC/TMD). They will be assessed in Visual analogue scale (VAS), sleep quality, Pressure Pain Threshold (PPT) and pressure pain tolerance (PPTol), and then allocated in one of the three interventions for 21 days: isometric mandibular active exercises over silicone bars; video-guided isotonic mandibular contractions over cloth pegs or counseling about disorders nature as passive comparison. After 21 days, VAS, PPT and PPTol in bilateral temporalis and masseter muscles will be assessed for a second time,) and compared with initial pain status.

Data will be entered by single blind operator, and will be open for quality auditing. Site monitoring will be performed by the University clinical entities.

Data checks will be also performed as planned. Descriptive and analytical statistics will be performed to address the primary and secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* Temporomandibular Myofascial pain diagnosis
* Oral contraceptives consumption
* Facial pain for at least 3 months (and at least 10 of the last 30 days at Visit 0)
* Agrees to terms for continuing/discontinuing certain prescription/over-the-counter pain medications.

Exclusion Criteria:

* Other orofacial pain diagnosis
* Oral surgery within 6 months
* Treatment for pain management within past 30 days
* Neurological or psychiatric disorders
* Orthodontic treatment
* History of pregnancy, pregnancy or breastfeeding.

Ages: 18 Years to 26 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2014-10-18 (Actual); Primary Completion 2016-12-06 (Actual); Study Completion 2016-12-30 (Actual)

PRIMARY OUTCOMES:
Change in the weekly mean subjective pain index after 21 days of treatment | Visit 1 (study day 0) and Visit 4 (study day 3) ( duration study 21 days)
  Weekly mean subjective pain computed as the arithmetic mean of daily pain subjective values (visual analog scale - VAS) in Visit 1and prior to each study visit. Daily pain index is computed as pain intensity (0-100 numeric rating scale where 0 = "no pain" and 100 = "the most intense pain imaginable") for the different muscular sites tested.
Change in the weekly mean pressure pain threshold (PPT) after 21 days of treatment | Visit 1 (study day 0) and Visit 4 (study day 3) ( duration study 21 days)
  Weekly mean pressure pain threshold is computed as the arithmetic mean of daily pressure pain threshold values for muscular sites in Visit 1and prior to each study visit. Pressure values, measured in kilogram-force (kgf), from up to 3 experimental pressure stimuli, bilaterally applied to the area of temporalis muscle, will be averaged to obtain a single pressure pain threshold value per anatomical site.
Change in the weekly mean pressure pain tolerance (PPTol) after 21 days of treatment | Visit 1 (study day 0) and Visit 4 (study day 3) ( duration study 21 days)
  Weekly mean pressure pain tolerance is computed as the arithmetic mean of daily pressure pain tolerance values for muscular sites in Visit 1and prior to each study visit. Plot is captured as a pressure value, measured in kilogram-force (kgf) in 1 experimental pressure stimuli, bilaterally applied per anatomical muscle site.

SECONDARY OUTCOMES:
Change in pressure pain threshold at temporalis muscle after 1 week of treatment | Visit 1 (study day 0) and Visit 2 (study day 7) ( 7 days in between)
  Pressure values, measured in kilogram-force (kgf), from up to 3 experimental pressure stimuli, bilaterally applied to the area of temporalis muscle, will be averaged to obtain a single pressure pain threshold value per anatomical site.
Change in pressure pain threshold at temporalis muscle after 2 weeks of treatment | Visit 1 (study day 0) and Visit 2 (study day 14) ( 7 days in between)
  Pressure values, measured in kilogram-force (kgf), from up to 3 experimental pressure stimuli, bilaterally applied to the area of temporalis muscle, will be averaged to obtain a single pressure pain threshold value per anatomical site.
Change in pressure pain threshold at temporalis muscle after 3 weeks of treatment | Visit 1 (study day 0) and Visit 2 (study day 21) ( 7 days in between)
  Pressure values, measured in kilogram-force (kgf), from up to 3 experimental pressure stimuli, bilaterally applied to the area of temporalis muscle, will be averaged to obtain a single pressure pain threshold value per anatomical site.
Change in pressure pain threshold at masseter muscle after 1 week of treatment | Visit 1 (study day 0) and Visit 2 (study day 7) ( 7 days in between)
  Pressure values, measured in kilogram-force (kgf), from up to 3 experimental pressure stimuli, bilaterally applied to the area of masseter muscle, will be averaged to obtain a single pressure pain threshold value per anatomical site.
Change in pressure pain threshold at masseter muscle after 2 weeks of treatment | Visit 1 (study day 0) and Visit 2 (study day 14) ( 14 days in between)
  Pressure values, measured in kilogram-force (kgf), from up to 3 experimental pressure stimuli, bilaterally applied to the area of masseter muscle, will be averaged to obtain a single pressure pain threshold value per anatomical site.
Change in pressure pain threshold at masseter muscle after 3 weeks of treatment | Visit 1 (study day 0) and Visit 2 (study day 21) ( 21 days in between)
  Pressure values, measured in kilogram-force (kgf), from up to 3 experimental pressure stimuli, bilaterally applied to the area of t masseter muscle, will be averaged to obtain a single pressure pain threshold value per anatomical site.
Change in pressure pain tolerance at temporalis muscle after 1 week of treatment | Visit 1 (study day 0) and Visit 2 (study day 7) ( 7 days in between)
  Pressure pain tolerance is captured as a pressure value, measured in kilogram-force (kgf) in 1 experimental pressure stimuli, bilaterally applied to the area of temporalis muscle.
Change in pressure pain tolerance at temporalis muscle after 2 weeks of treatment | Visit 1 (study day 0) and Visit 2 (study day 14) ( 14 days in between)
  Pressure pain tolerance is captured as a pressure value, measured in kilogram-force (kgf) in 1 experimental pressure stimuli, bilaterally applied to the area of temporalis muscle.
Change in pressure pain tolerance at temporalis muscle after 3 weeks of treatment | Visit 1 (study day 0) and Visit 2 (study day 21) ( 21 days in between)
  Pressure pain tolerance is captured as a pressure value, measured in kilogram-force (kgf) in 1 experimental pressure stimuli, bilaterally applied to the area of temporalis muscle.
Change in pressure pain tolerance at masseter muscle after 1 week of treatment | Visit 1 (study day 0) and Visit 2 (study day 7) ( 7 days in between)
  Pressure pain tolerance is captured as a pressure value, measured in kilogram-force (kgf) in 1 experimental pressure stimuli, bilaterally applied to the area of masseter muscle.
Change in pressure pain tolerance at masseter muscle after 2 weeks of treatment | Visit 1 (study day 0) and Visit 2 (study day 14) ( 14 days in between)
  Pressure pain tolerance is captured as a pressure value, measured in kilogram-force (kgf) in 1 experimental pressure stimuli, bilaterally applied to the area of masseter muscle.
Change in pressure pain tolerance at masseter muscle after 3 weeks of treatment | Visit 1 (study day 0) and Visit 2 (study day 21) ( 21 days in between)
  Pressure pain tolerance is captured as a pressure value, measured in kilogram-force (kgf) in 1 experimental pressure stimuli, bilaterally applied to the area of masseter muscle.
Change in the Pittsburgh Sleep Quality Index (PSQI) global score after 21 days of treatment | Visit 1 (study day 0) and Visit 4 (study day 3) ( duration study 21 days)
  The PSQI has 19 items grouped into 7 component scores, each weighted equally on a 0-3 scale. The 7 component scores are summed to obtain a global score, which has a range of 0-21.

CONTACTS AND LOCATIONS:
Overall Officials: Juan F Oyarzo, Prof, Principal Investigator — Universidad Andres Bello

IPD SHARING:
Plan to Share IPD: No
no plan